CLINICAL TRIAL: NCT01291160
Title: A Prospective, Randomized Blinded Multicenter, Parallel Study Comparing Transdermal, Continuous Oxygen Delivery to Moist Wound Therapy (MWT) in the Treatment of Diabetic Foot Ulcers
Brief Title: Transdermal Continuous Oxygen Therapy for Diabetic Foot Ulcers
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Neogenix, LLC dba Ogenix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EPF-409
Record Dates: First submitted 2011-02-04; First posted 2011-02-08 (Estimated); Results first posted 2014-05-13 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-04

CONDITIONS: Diabetic Foot Ulcers
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Epiflo Treatment (Experimental): The cohort will comprise of 2 populations: the Treatment Arm of up to 90 subjects; and the Control Arm of up to 90 subjects, in order to collect 120 invaluable subjects. The Treatment Arm includes subjects with DFU who will receive EPIFLO in addition to standard wound care therapy during the Treatment Period.
  Interventions: Device: Epiflo
- Sham Device (Sham Comparator): The cohort will comprise of 2 populations: the Treatment Arm of up to 90 subjects; and the Control Arm of up to 90 subjects, in order to collect 120 invaluable subjects. Control Arm includes subjects with Diabetic Foot Ulcers who will receive sham units of EPIFLO along with standard wound care therapy during the treatment Period.
  Interventions: Other: Moist Wound Therapy

INTERVENTIONS:
Device: Epiflo — During the Treatment Period, subjects will be administered EPIFLO (either working units or sham units per randomization schedule) in conjunction with standard wound therapy regimen consisting of aggressive debridement, wound cleansing, wound dressing, for a period of 12 weeks, or until the wound completely closes, whichever event occurs first.
  Other Names: Transdermal Continuous Oxygen Therapy
  Arms: Epiflo Treatment
Other: Moist Wound Therapy — During the Treatment Period, subjects will be administered EPIFLO (either working units or sham units per randomization schedule) in conjunction with standard wound therapy regimen consisting of aggressive debridement, wound cleansing, wound dressing, for a period of 12 weeks, or until the wound completely closes, whichever event occurs first.
  Arms: Sham Device

SUMMARY:
This is a multicenter, prospective, parallel, double-blinded, validation study of up to 12 weeks duration to evaluate the safety and effectiveness of EPIFLO for the treatment of Diabetic Foot Ulcer. The primary objectives of this study are: 1) to evaluate the effectiveness of EPIFLO in combination with standard wound therapy on wound healing as compared to standard wound therapy alone; and 2) Screening for potential safety issues.

Diabetic subjects with a Diabetic Foot Ulcer present for a minimum of 30 days will be enrolled. All subjects enrolled in the study will receive a standard wound therapy regimen consisting of, wound cleansing, moist wound care, off-loading and as appropriate, aggressive debridement. Subjects will be randomized to either the Treatment arm or the Control arm. Subjects will be assessed weekly for signs of wound healing during the 12-week Treatment Period, once two weeks after wound closure and once at the end of 12-week durability Period.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 20-90 years of age with type 1 or type 2 diabetes mellitus with non-healing, full-thickness, University of Texas Classification of Diabetic Foot Ulcers Class IA diabetic foot ulcers of at least 4 weeks duration, but not greater than 52 weeks, measuring 1 -10 cm2 in area (Area = length x width) 50% at least from 65+ age group
* Any diabetic foot ulcer at or below the malleoli
* Patients with partial amputation up to & including a TMA
* Subjects; between 20-90 years of age with a diabetic foot ulcer; 50% at least from 65+ age group
* Subjects must have had the wound open for at least 4 weeks from day one on screening visit.
* Subjects wound must be ≥1 cm2 in size at screening visit, but not greater than 10 cm2.
* Subject's ABI should be ≥ 0.7 on the study limb or transcutaneous partial pressure oxygen (TcpO2) >40mmHg; or a toe pressure ≥40mmHg; or a Doppler waveform consistent with adequate flow in the foot(biphasic or triphasic waveforms) at screening
* No active malignancy except non-melanoma skin cancer
* Subject and/or caregiver must be willing and able to learn and perform the duties of dressing changes, and demonstrate the ability to do so.
* If patient has had a history of alcohol or substance abuse within 6 months prior to base line period, should provide proof of treatment.

Exclusion Criteria:

* Wounds of duration >52 weeks
* Evidence of gangrene on any part of affected limb;
* Subjects with active Charcot's foot on the study limb;
* Subjects scheduled to undergo vascular surgery, angioplasty or thrombolysis;
* Subjects with infected target ulcers, accompanied by cellulitis, known or suspected osteomyelitis, or other clinical evidence of infection;
* Index ulcer has exposed tendons, ligaments, muscle, or bone.
* ulcers present in between toes
* Target limb is infected at beginning of study
* Must never have had malignancy on study limb
* Oral, or IV antibiotic/antimicrobial agents or medications have been used within 2 days (48 hours) of baseline.
* Patients with steroids >7mg dosage are excluded
* Subject has received growth factor therapy (e.g., autologous platelet-rich plasma gel, becaplermin, bilayered cell therapy, dermal substitute, extracellular matrix) within two weeks of screening date.
* Subject may not be pregnant at the time of treatment.
* Subjects with ulcer that has a total Surface Area of greater than 10 cm2 at Screening Visit as measured by a member of the study staff;
* Subject is undergoing renal dialysis, has known immune insufficiency, other than Diabetes Mellitus
* Ulcers which decrease in area by >30% during the screening 1-week run-in period
* History of peripheral vascular repair within the 30 days of baseline.
* Subject is currently receiving or has received radiation or chemotherapy within 3 months of randomization.
* No known "patient-reported" alcohol or substance abuse within three months prior to baseline.
* Subject currently enrolled or participated within 30 days of baseline in another investigational device, drug or biological trial.
* Subject allergic to a broad spectrum of primary & secondary dressing materials,including occlusive dressings and the adhesives on such dressings.
* Subject with Chopart amputation

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2009-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vickie R Driver, MSDPM FACFAS, Principal Investigator — Lead Principal Investigator
Locations (14):
- United States (14):
  - Carl T. Hayden VA Medical Center, Phoenix, Arizona
  - Southern AZ VA Health Care System, Tucson, Arizona
  - Dean Vayser, DPM, Encinitas, California
  - California School of Podiatric Medicine, Fresno, California
  - Los Angeles, California
  - San Jose, California
  - The Diabetic Foot, San Marcos, California
  - UF College of Medicine-Jacksonville, Jacksonville, Florida
  - Bruce W. Carter Dept. of Veterans Affairs Medical Center, Miami VA Health Care System, Miami, Florida
  - Boston Medical Center, Boston, Massachusetts
  - Ocean County Foot & Ankle Surgical Associates, Toms River, New Jersey
  - Ohio College of Podiatric Medicine, Independence, Ohio
  - San Antonio, Texas
  - Tacoma Diabetic Foot Center, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Epiflo Treatment | Sham Device
Started | 66 | 64
Completed | 48 | 48
Not Completed | 18 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Epiflo Treatment | Sham Device | Total
Number analyzed (Participants) | 66 | 64 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.25 (13.06) | 58.46 (9.53) | 59.25 (13.06)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 47 | 94
  >=65 years | 19 | 17 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 15 | 36
  Male | 45 | 49 | 94

OUTCOME MEASURES:

1. Primary Outcome: Number of 100% Wound Closure
Time Frame: before or at week 12
Population: Analyzed the per-protocol population
Measure: Number; unit: percentage of patients
Arm/Group | Epiflo Treatment | Sham Device
Number analyzed (Participants) | 61 | 61
percentage of patients | 55.74 | 50.82

ADVERSE EVENTS:
Arm/Group | Epiflo Treatment | Sham Device
Serious Adverse Events (participants affected / at risk) | 10/66 | 9/64
Other Adverse Events (participants affected / at risk) | 37/66 | 37/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epiflo Treatment (N=66) | Sham Device (N=64)
Cellulitis (Infections and infestations) | 1 (1) | 3 (3) — Cellulitis of leg
Wound Infection (Infections and infestations) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Gas gangrene (Infections and infestations) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epiflo Treatment (N=66) | Sham Device (N=64)
Abrasions (Injury, poisoning and procedural complications) | 2 (2) | 5 (6)
Cellulitis (Infections and infestations) | 1 (1) | 3 (3)
Diabetic ulcer (Vascular disorders) | 5 (8) | 3 (3)
Edema (General disorders) | 1 (2) | 4 (4)
Wound Infection (Infections and infestations) | 2 (2) | 3 (3)
Wound complication (Injury, poisoning and procedural complications) | 30 (52) | 32 (55)
Wound infection (Infections and infestations) | 3 (3) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No